CLINICAL TRIAL: NCT00170924
Title: A Multi-center, Randomized, Placebo-controlled, Double-blind Study to Evaluate the Effect of the Angiotensin II Antagonist Valsartan on Diastolic Function in Patients With Hypertension and Diastolic Dysfunction
Brief Title: To Find Out Whether Valsartan With or Without Other Blood Pressure Medications Would Improve the Ability of the Heart to Fill and Empty, and the Ability of the Heart Muscle to Relax Adequately in People With High Blood Pressure.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CVAL489AUS52
Record Dates: First submitted 2005-09-10; First posted 2005-09-15 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2011-11

CONDITIONS: Diastolic Dysfunction; Hypertension
Keywords: Hypertension, High Blood Pressure, Diastolic Dysfunction,; Heart Disease
MeSH Terms: conditions — Hypertension; Heart Diseases | interventions — Valsartan

INTERVENTIONS:
Drug: Valsartan

SUMMARY:
Patients who have had high blood pressure for a long time may have diastolic dysfunction. Diastolic Dysfunction is when your heart has difficulty filling and emptying, and relaxing adequately.

This study is to find out if Valsartan) will improve the ability of the heart to fill, empty, and relax appropriately when given alone or with other medicines to treat high blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis/History of high blood pressure
* Male or Female age 45 years or older

Exclusion Criteria:

* History of stroke, transient ischemic attack or heart attack within the last 6 months
* A hospital admission for congestive heart failure within the last year
* Use of certain high blood pressure medications such as ACE inhibitors, Angiotensin Receptor Blockers or aldosterone antagonists or other agents that may work in the same pathway (RAAS) as valsartan within the past 3 months.

Other protocol-defined exclusion criteria may apply.

Min Age: 45 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 317 (Actual)
Dates: Start 2004-08; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in diastolic heart function at 38 weeks, measured by echocardiogram

SECONDARY OUTCOMES:
Change from baseline in the wall thickness of left heart ventricle after 38 weeks
Change from baseline in the size (mass) left heart ventricle after 38 weeks
Change from baseline in heart function after 38 weeks
Change from baseline in circulating marker of ventricular function after 38 weeks
Change from baseline in circulating marker of inflammation

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States

REFERENCES:
- [Derived] Solomon SD, Janardhanan R, Verma A, Bourgoun M, Daley WL, Purkayastha D, Lacourciere Y, Hippler SE, Fields H, Naqvi TZ, Mulvagh SL, Arnold JM, Thomas JD, Zile MR, Aurigemma GP; Valsartan In Diastolic Dysfunction (VALIDD) Investigators. Effect of angiotensin receptor blockade and antihypertensive drugs on diastolic function in patients with hypertension and diastolic dysfunction: a randomised trial. Lancet. 2007 Jun 23;369(9579):2079-87. doi: 10.1016/S0140-6736(07)60980-5. PMID 17586303
- See also: Novartis Patient Recruitment Website — http://www.novartisclinicaltrials.com